CLINICAL TRIAL: NCT01116700
Title: The Pharmacokinetics and Pharmacodynamics of Dexmedetomidine in Patients With Seizure Disorders
Brief Title: Dexmedetomidine in Seizure Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UCSF-AF-02-2010
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Seizure Disorders
Keywords: Epilepsy; Dexmedetomidine; Seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be administered to 2 groups: (1) Seizure disordered patients on anticonvulsants and (2) Healthy volunteers (Control group)
  Other Names: Precedex

SUMMARY:
Dexmedetomidine is an alpha-2 agonist commonly used during neurosurgery due to its unique properties as a sedative and anxiolytic with minimal respiratory depression. Neurosurgical patients frequently come to the operating room on anticonvulsant therapy with a history of seizures. The investigators clinical experience suggests that these patients are resistant to the sedative effects of dexmedetomidine. This effect may represent a pharmacokinetic interaction between the anticonvulsant medications and dexmedetomidine or the higher dexmedetomidine dose requirement could result from abnormal pharmacodynamics due to the underlying seizure disorder. The investigators study aims to investigate the pharmacokinetic and pharmacodynamic differences of dexmedetomidine between patients receiving and not receiving enzyme-inducing anticonvulsant therapy and to identify a potential mechanism for these differences.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, BMI 20-25 kg/m2
* Anticonvulsant Group: Diagnosis of seizure disorder taking carbamazepine or phenytoin for a minimum of 2 weeks
* Control Group: Healthy volunteers taking no medications

Exclusion Criteria:

* Positive urine pregnancy test or lactating
* History of allergy to dexmedetomidine or alpha -2 agonists
* History of liver, renal or thyroid disease
* History of cardiovascular disease including history of arrhythmia or congestive heart failure
* History of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Serum level of dexmedetomidine | 0-8 hour period
  Serum levels of dexmedetomidine will be taken at specific intervals during and after a step-wise computer controlled infusion of dexmedetomidine.

SECONDARY OUTCOMES:
Patient State Index (PSI) and Entropy | 0-8h
  PSI and/or state entropy will be recorded at specific intervals during and after a step-wise computer controlled infusion of dexmedetomidine.
Visual Analog Scale score | 0-8h
  VAS scores will be recorded at specific intervals during and after a step-wise computer controlled infusion of dexmedetomidine.
Ramsay Sedation Score | 0-8h
  Ramsay sedation scores will be recorded at specific intervals during and after a step-wise computer controlled infusion of dexmedetomidine.
Observer's Assessment of Alertness/Sedation Score (OAA/S) | 0-8h
  OAA/S scores will be recorded at specific intervals during and after a step-wise computer controlled infusion of dexmedetomidine.

CONTACTS AND LOCATIONS:
Overall Officials: Alana M Flexman, MD, Principal Investigator — UCSF Department of Anesthesia; Pekka Talke, MD, Principal Investigator — UCSF Department of Anesthesia; Paul Garcia, MD, Principal Investigator — UCSF Department of Neurology
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Sleigh JW, Vacas S, Flexman AM, Talke PO. Electroencephalographic Arousal Patterns Under Dexmedetomidine Sedation. Anesth Analg. 2018 Oct;127(4):951-959. doi: 10.1213/ANE.0000000000003590. PMID 29933272